CLINICAL TRIAL: NCT03432702
Title: Horizontal Ridge Augmentation With Guided Bone Regeneration Using Particulate Xenogenic Bone Substitutes With or Without Autogenous Block Grafts: A Randomized Controlled Trial
Brief Title: Horizontal Ridge Augmentation With or Without Autogenous Block Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Científica del Sur (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00013
Record Dates: First submitted 2018-01-31; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Bone Regeneration; Bone Transplantation; Bone Substitutes; Cone-beam Computed Tomography; Dental Implants
MeSH Terms: interventions — Alveolar Ridge Augmentation; Bone Transplantation

STUDY DESIGN:
Intervention Model Description: Single center, prospective, controlled, parallel-armed, randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome measurements will be recorded by an examiner, who will not participate in any study procedure, and will be blind to the allocated treatment. This blinded examiner will be trained and calibrated to perform measurements. A dentist who is blinded to the treatment protocol will performe all radiographic measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alveolar ridge augmentation without ABG (Active Comparator): Horizontal ridge augmentation using guided bone regeneration without autogenous block graft (ABG)
  Interventions: Procedure: Horizontal ridge augmentation
- Alveolar ridge augmentation with ABG (Experimental): Horizontal ridge augmentation using guided bone regeneration with autogenous block graft (ABG).
  Interventions: Procedure: Horizontal ridge augmentation

INTERVENTIONS:
Procedure: Horizontal ridge augmentation — Surgical procedures performed to provide the alveolar ridge with enough width and height to allow for the prosthetically driven implant placement.
  Other Names: Alveolar ridge augmentation; Bone grafting

SUMMARY:
To evaluate dimensional bone alterations following horizontal ridge augmentation using guided bone regeneration (GBR) with or without autogenous block graft (ABG) for the rehabilitation of atrophic jaws with dental implants.

DETAILED DESCRIPTION:
Forty-two patients with 42 severe horizontal bone atrophy sites in the maxilla or mandible will be randomly assigned to two groups: ABG or GBR.

In the ABG group, a combination of ABG with particulate xenograft, covered with collagen membrane, will be used, while only a combination of particulate xenograft and collagen membrane alone will be in the GBR group. After 6-9 months of healing, implants were inserted. All implants will be definitively restored 6 months after implant placement. Radiographic examination (cone beam computed tomograms, CBCT) will be performed to evaluate the amount of horizontal bone width (HBW) gain immediately after bone grafting procedure (T0), at 6 months (T6), and at 18 months (T18). Patient demographic information, amount of width augmentation, implant survival, complications, and contributing factors will be gathered and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old, who required an implant supported restoration in at least one site, with severe atrophy of the alveolar ridge in the horizontal plane (class III-IV atrophy according to Cawood and Howell classification),
* adequate oral hygiene
* no history of previous bone augmentation procedures at the implant site, and
* able to understand and sign an informed consent form.

Exclusion Criteria:

* uncontrolled systemic conditions, irradiation in the head and neck area, - immunosuppressed or immunocompromised,
* presented with oral disorders (such as lichen planus),
* treated or under treatment with intravenous amino-bisphosphonates,
* untreated periodontitis, poor oral hygiene and motivation,
* parafunctional habits,
* pregnant or lactating,
* drug or alcohol abuse,
* psychiatric disorders,
* a history (within the last 3 months) of using (at least weekly or more frequently) smokeless chewing tobacco, smoking a pipe, cigar or cigarette (at a rate of more than 10 cigarettes per day),
* acute/chronic infection/inflammation in the area, or
* an extraction with less than 3 months of healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in horizontal alveolar ridge width from pre-operatively (baseline) to 12 months after implant loading. | From pre-operatively (baseline) to 12 months after implant loading.
  Horizontal alveolar ridge changes in being assessed in the regenerated area. This outcome will be evaluated from pre-operatively (baseline), to 12 months after implant loading by measuring the alveolar ridge width at various points on the cross-sectional images using data obtained from CBCT scans.

SECONDARY OUTCOMES:
Implant failure | At 6 months (T6), and at 18 months (T18) after implant placement.
  The presence of an implant that requires implant removal (e.g., implant mobility).
Complications | 6 months
  Assessments of complications related to study procedures will be recorded during the follow up period.
Regrafting necessity | At 6 months (T6).
  Number of implants that needed regrafting to allow for ideal prosthetically driven implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Mendoza-Azpur, DDS, Principal Investigator — Científica del Sur University
Locations (1):
- Periodontal Postgraduate Clinic at the Faculty of Dentistry, Científica del Sur University, Lima, Peru

IPD SHARING:
Plan to Share IPD: No